CLINICAL TRIAL: NCT05719493
Title: Effectiveness and Health Benefits of a Nutritional, Chronobiological and Physical Exercise Primary Care Intervention in Fibromyalgia and Chronic Fatigue Syndrome: SYNCHRONIZE + Mixed Methods Study Protocol.
Brief Title: Effectiveness and Health Benefits of a Nutritional, Chronobiological and Physical Exercise Intervention in Fibromyalgia and Chronic Fatigue Syndrome (SYNCHRONIZE +)
Acronym: SYNCHRONIZE +
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: SLT/21/000009
Record Dates: First submitted 2023-01-30; First posted 2023-02-09 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Fibromyalgia; Chronic Fatigue Syndrome
Keywords: multicomponent intervention; nutrition; chronobiology; physical exercise; quality of life; primary health care
MeSH Terms: conditions — Fibromyalgia; Fatigue Syndrome, Chronic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- multicomponent-treatment no benefiting group (No Intervention): Participants in the control group will receive the care from the usual clinical practice
- munticomponent-treatment benefiting group (Experimental): Partcipants in the intervention group will receive the care from the usual practice plus the studied intervention.
  Interventions: Other: multicomponent treatment

INTERVENTIONS:
Other: multicomponent treatment — The intervention to be evaluated consists of 4 group sessions carried out in two weeks, 6 hours per week divided in 2 days (a total of 12 hours), of active education in nutrition, chronobiology and physical exercise in people diagnosed with Chronic Fatigue Syndrome and Fibromyalgia.
  Arms: munticomponent-treatment benefiting group

SUMMARY:
Chronic pain, fatigue and insomnia are classical symptoms of Fibromyalgia and Chronic Fatigue Syndrome, affecting seriously life quality. Non-pharmacological multicomponent approach is gaining relevance in Fibromyalgia treatment. However, nutrition and chronobiology are often not approached in-depth despite their potential. Furthermore, programs addressed to Chronic Fatigue Syndrome are still scare. This study aims to evaluate the effectiveness of a compact multidisciplinary group intervention based on nutrition, chronobiology and physical exercise in the improvement of lifestyle and life quality in Fibromyalgia and Chronic Fatigue syndrome.

DETAILED DESCRIPTION:
The investigators will perform a mixed study through a randomized clinical trial in Catalonian Primary Care with patients diagnosed of Fibromyalgia (M79.7) or both Fibromyalgia and Chronic Fatigue Syndrome (G93.3). The control group will follow the usual clinical practice and the intervention group, the usual practice plus the studied intervention (12 hours in 4 days). The intervention (based on nutrition, chronobiology and physical exercise) will be designed taking into account participant's opinion through focus groups. In both groups, quality of life (EuroQol-5D), as well as MFI, VAS pain, PSQI, erMEDAS-17, BRIAN, REGICOR-Short, FIQR and HADs questionnaires will be collected, prior to the intervention, and 1, 3, 6 and 12 months post-intervention. Food intake, body composition, resistance and strength will also be evaluated. The effect size will be calculated using Cohen's d and logistic regression models will be used to quantify the impact of the intervention by adjusting for different variables. In addition, a qualitative analysis with a descriptive phenomenological perspective from post-intervention focus groups of participants and professionals will be done.

ELIGIBILITY:
Inclusion Criteria:

* People aged 18-65, recent diagnosis of Fibromyalgia (M79.1) (<10 years), or diagnosis of Fibromyalgia and Chronic Fatigue Syndrome (M79 .7 and G93.3), with availability, motivation and interest in the intervention.

Exclusion Criteria:

* not meeting the inclusion criteria, being participating in other group interventions aimed at the treatment of these syndromes, presence of severe mental comorbidity or other relevant medical disorders or pathologies that may interfere with the evaluation of the intervention

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2021-10-04 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
change in quality of life | change from life quality at 1, 3, 6 and 12 months after the beginning of the intervention
  to be evaluated with the EuroQol-5D questionnaire. It will be measured by a scale Likert: 0 (worst health) to 100 (better health) and a descriptive system with five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression; with five levels of severity in each dimension: no problems, mild problems, moderate problems, severe problems, and extreme problems/impossibility.

SECONDARY OUTCOMES:
change in fatigue indicator | change from fatigue indicator at 1, 3, 6 and 12 months after the beginning of the intervention
  to be evaluated with the "Multidimensional Fatigue Inventory" (MFI) questionnaire (Smet et al., 1995). It will measure 20-items. MFI-20 has an even proportion of positively and negatively worded items that are rated on a 5-point Likert scale. Subscale scores (range 4-20) are calculated as the sum of item ratings and a total fatigue score (range 20-100) is calculated as the sum of subscale scores. Higher scores indicate a higher level of fatigue.
change in sleep quality and insomnia indicator | change from sleep quality and insomnia indicator at 1, 3, 6 and 12 months after the beginning of the intervention
  Sleep quality and insomnia will be assessed with the Pittsburgh Sleep Quality Index (PSQI-19 items) (Buysse et al., 1989). In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
change in pain indicator | change from pain indicator at 1, 3, 6 and 12 months after the beginning of the intervention
  To assess pain, the VAS questionnaire will be used (Marques et al., 2008). It will be measured by a scale Likert: 0 (absence of pain) to 10 (worst possible pain).
change in adherence to the Mediterranean diet | change from adherence to the Mediterranean diet at 1, 3, 6 and 12 months after the beginning of the intervention
  adherence to the Mediterranean diet will be assessed with the erMEDAS-17-item questionnaire (PREDIMED Plus; Schröder et al., 2021). Adherence to dietary habits characteristic of a MedDiet is scored, in each item, with 1 point and the opposite, with 0 points. Total scoring scale goes from 0 to 17 points, where 0 means no adherence and 17, maximum adherence. The score can be also classified into approximate tertiles: low (≤ 7), medium (8-10), and high (11-17).
change in physical exercise practice and sedentary lifestyle | change from physical exercise practice and sedentary lifestyle at 1, 3, 6 and 12 months after the beginning of the intervention
  physical exercise practice and sedentary lifestyle will be assessed with the REGICOR-Short questionnaire (Molina et al., 2017). The short questionnaire estimates energy expenditure in total physical activity and by intensity (light, moderate, vigorous) following REGICOR-Short algoritmes, and includes 2 questions about sedentary behavior and a question about occupational physical activity. We will evaluate change in amount of time dedicated to physical activity (minutes or hours) and physical activity intensity per week (energy expenditure or METs x min/week), and change in sedentarism (number of hours per week doing sedentary activities).
change in circadian biological rhythm | change from circadian biological rhythm at 1, 3, 6 and 12 months after the beginning of the intervention
  the circadian biological rhythm will be assessed with the "Biological Rhythms Interview of Assessment in Neuropsychiatry" (BRIAN) questionnaire (Giglio et al., 2008). The BRIAN includes 18-items to investigate four main areas related to circadian rhythm disturbance: sleep, activities, social rhythms and eating patterns. Items are rated using a 4-point scale, (1)= no difficulty, (2)= mild difficulty, (3)= moderate difficulty, and (4) =severe difficulty. The BRIAN scores thus range from 1 to 72, where the higher scores suggest severe circadian rhythm disturbance.
change in functional impact of fibromyalgia | change from functional impact of fibromyalgia at 1, 3, 6 and 12 months after the beginning of the intervention
  to be evaluatedwith the Revised Questionnaire on the Impact of Fibromyalgia (FIQR). It will be measured by a scale Likert: 0 (best) to 100 (worst).
change in mood indicator (anxiety) | change from mood indicator (anxiety) at 1, 3, 6 and 12 months after the beginning of the intervention
  To be evaluated with the Hospital Anxiety and Depression Scale (HADS) questionnaire. The scale llikert punctuates from 0 to 21 (8 to 10 indicates a doubtful case of anxiety; more than 11 indicates a probable case of anxiety)
change in food intake | change from food intake at at 1, 3, 6 and 12 months after the beginning of the intervention
  Will be evaluate through R24h and FFQ (Rodríguez et al., 2008). The R24h will be evaluated qualitatively (number of intakes/day; intake composition, etc.) while the FFQ register weekly and monthly intake of different food (times per week; times per month), and will evaluated qualitatively.
change in body mass index (BMI) | change from BMI at 1, 3, 6 and 12 months after the beginning of the intervention
  Weight and height will be combined to report BMI in Kg/m2.
change in body fat | change from body fat at 1, 3, 6 and 12 months after the beginning of the intervention
  Body fat (measured in %) will be measured by bioimpedance with a OMRON BF511 body composition monitor.
change in skeletal muscle | change from skeletal muscle at 1, 3, 6 and 12 months after the beginning of the intervention
  Skeletal muscle (measured in %) will be measured by bioimpedance with a OMRON BF511 body composition monitor.
change in endurance | change from endurance at 1, 3, 6 and 12 months after the beginning of the intervention
  Endurance will be evaluated with the ''6-min walk test' (Rikli and Jones, 1999). This test involves determining the maximum distance (m) that can be walked in 6 min .
change in lower body muscular strength | change from lower body muscular strength at 1, 3, 6 and 12 months after the beginning of the intervention
  The ''30-s chair stand test''(Rikli and Jones, 1999) involves counting the number of times within 30 s that an individual can rise to a full stand from a seated position with the back straight and the feet flat on the floor, without pushing off with the arms.
change in upper body muscular strength | change from upper body muscular strength at at 1, 3, 6 and 12 months after the beginning of the intervention
  The handgrip strength will be assessed using a "hand dynamometer". The subject continuously and gradually squeezes for at least 2 s. Each patient completes two attempts with each hand, with the arm fully extended, forming an angle of 30- with respect to the trunk. The maximum score in kilograms for each hand is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Català de la Salut, Tortosa, Tarragona, Spain